CLINICAL TRIAL: NCT00923702
Title: Randomised Trial of Two Versus Three Doses of Human Papillomavirus (HPV) Vaccine in India
Brief Title: Trial of Two Versus Three Doses of Human Papillomavirus (HPV) Vaccine in India
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Partha Basu (Other)
Collaborators: All India Institute of Medical Sciences (Other); Cancer Foundation of India (Other); Christian Fellowship Community Health Centre (Other); German Cancer Research Center (Other); Gujarat Cancer & Research Institute (Other); Jehangir Clinical Development Centre (Other); MNJ Institute of Oncology and Regional Cancer Center (Other Government); Rajiv Gandhi Centre for Biotechnology (Industry); Nargis Datta Memorial Cancer Hospital (Other); Tata Memorial Centre (Other)
Responsible Party: Sponsor-Investigator, Partha Basu, Early Detection, Prevention and Infection Branch at IARC, WHO, International Agency for Research on Cancer
Organization: International Agency for Research on Cancer (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BMGF48979; ISRCTN98283094 (Other: BioMedCentral); REFCTRI-2009 000137 (Registry Identifier: Indian Clinical Trial Registry)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2022-10-20 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer; Cervical Precancerous Lesions
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 3-dose (Active Comparator): The participants received three doses of the Prophylactic quadrivalent HPV vaccine Merck (Gardasil®) at days 1, 60 and 180+.
  Interventions: Biological: Prophylactic quadrivalent HPV vaccine Merck (Gardasil®)
- 2-dose (Experimental): The participants received two doses of the Prophylactic quadrivalent HPV vaccine Merck (Gardasil®) at days 1 and 180+.
  Interventions: Biological: Prophylactic quadrivalent HPV vaccine Merck (Gardasil®)
- 2 doses by default (Experimental): The participants received two doses of the Prophylactic quadrivalent HPV vaccine Merck (Gardasil®) at days 1 and 60 by default (incomplete doses)
  Interventions: Biological: Prophylactic quadrivalent HPV vaccine Merck (Gardasil®)
- Single-dose (Experimental): The participants received one dose of the Prophylactic quadrivalent HPV vaccine Merck (Gardasil®) by default (incomplete doses)
  Interventions: Biological: Prophylactic quadrivalent HPV vaccine Merck (Gardasil®)
- Unvaccinated (No Intervention): A cohort of unvaccinated women

INTERVENTIONS:
Biological: Prophylactic quadrivalent HPV vaccine Merck (Gardasil®) — The participants received either one, two or three doses of the avaccine. Each injection contains 20 microgram type 6, 40 microgram type 11, 40 microgram type 16, and 20 microgram type 18.
  Other Names: Gardasil®
  Arms: 2 doses by default; 2-dose; 3-dose; Single-dose

SUMMARY:
The primary study hypothesis wasthat a two-dose human papillomavirus (HPV) vaccine regimen would offer similar immunogenicity and protection as that of a three-dose regimen to girls against persistent HPV infection and cervical neoplasia caused by HPV types included in the vaccine. The Government of India stopped vaccination in all the HPV vaccine trials in the country in April 2010 due to reasons not related to this study.

DETAILED DESCRIPTION:
The suspension of vaccination resulted in girls receiving 3 doses (days 1, 60 and ≥180), receiving 2 doses (days 1 and ≥180), receiving 2 doses at days 1 and 60 due to incomplete treatment ("by default"), and receiving one dose by default. A first age and site-matched cohort of unvaccinated married women was recruited, starting in May 2012 to serve as the unvaccinated control group of women for the analysis of HPV incidence and persistence outcomes. A second age and site-matched (age and site matched to the vaccinated women undergoing screening) cohort of unvaccinated married women is being recruited starting in June 2017 and is to be used in addition to the first unvaccinated cohort for the assessment of the cervical neoplasia outcome.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy, ambulant girls aged 10 - 18 years
* Unmarried girls
* Girls with intact uterus
* Resident in the villages chosen for the study

Exclusion Criteria:

* Girls with any severe and/or debilitating illness
* Past history of allergy to any medication

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22729 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Partha Basu, MD, Principal Investigator — International Agency for Research on Cancer
Locations (8):
- India (8):
  - MNJ Institute of Oncology & Regional Cancer Center, Hyderabad, Andhra Pradesh
  - Gujarat Cancer & Research Institute (GCRI), Ahmedabad, Gujarat
  - Tata Memorial Centre Rural Cancer Project, Nargis Dutt Memorial Cancer Hospital, Barshi, Maharashtra
  - Tata Memorial Center, Tata Memorial Hospital & Cancer Research Inst, Mumbai, Maharashtra
  - Jehangir Clinical Development Centre (JCDC) Pvt. Ltd., Pune, Maharashtra
  - Christian Fellowship Community Health Centre, Ambilikkai, Tamil Nadu
  - Cancer Foundation of India, Kolkata, West Bengal
  - All India Institute of Medical Sciences, New Delhi

REFERENCES:
- [Background] Basu P, Malvi SG, Joshi S, Bhatla N, Muwonge R, Lucas E, Verma Y, Esmy PO, Poli URR, Shah A, Zomawia E, Pimple S, Jayant K, Hingmire S, Chiwate A, Divate U, Vashist S, Mishra G, Jadhav R, Siddiqi M, Sankaran S, Prabhu PR, Kannan TPRA, Varghese R, Shastri SS, Anantharaman D, Gheit T, Tommasino M, Sauvaget C, Pillai MR, Sankaranarayanan R. Vaccine efficacy against persistent human papillomavirus (HPV) 16/18 infection at 10 years after one, two, and three doses of quadrivalent HPV vaccine in girls in India: a multicentre, prospective, cohort study. Lancet Oncol. 2021 Nov;22(11):1518-1529. doi: 10.1016/S1470-2045(21)00453-8. Epub 2021 Oct 8. PMID 34634254
- [Result] Sankaranarayanan R, Prabhu PR, Pawlita M, Gheit T, Bhatla N, Muwonge R, Nene BM, Esmy PO, Joshi S, Poli UR, Jivarajani P, Verma Y, Zomawia E, Siddiqi M, Shastri SS, Jayant K, Malvi SG, Lucas E, Michel A, Butt J, Vijayamma JM, Sankaran S, Kannan TP, Varghese R, Divate U, Thomas S, Joshi G, Willhauck-Fleckenstein M, Waterboer T, Muller M, Sehr P, Hingmire S, Kriplani A, Mishra G, Pimple S, Jadhav R, Sauvaget C, Tommasino M, Pillai MR; Indian HPV Vaccine Study Group. Immunogenicity and HPV infection after one, two, and three doses of quadrivalent HPV vaccine in girls in India: a multicentre prospective cohort study. Lancet Oncol. 2016 Jan;17(1):67-77. doi: 10.1016/S1470-2045(15)00414-3. Epub 2015 Dec 2. PMID 26652797
- [Result] Sankaranarayanan R, Joshi S, Muwonge R, Esmy PO, Basu P, Prabhu P, Bhatla N, Nene BM, Shaw J, Poli URR, Verma Y, Zomawia E, Pimple S, Tommasino M, Pawlita M, Gheit T, Waterboer T, Sehr P, Pillai MR; Indian HPV vaccine study group. Can a single dose of human papillomavirus (HPV) vaccine prevent cervical cancer? Early findings from an Indian study. Vaccine. 2018 Aug 6;36(32 Pt A):4783-4791. doi: 10.1016/j.vaccine.2018.02.087. Epub 2018 Mar 15. PMID 29551226
- [Result] Bhatla N, Nene BM, Joshi S, Esmy PO, Poli URR, Joshi G, Verma Y, Zomawia E, Pimple S, Prabhu PR, Basu P, Muwonge R, Hingmire S, Sauvaget C, Lucas E, Pawlita M, Gheit T, Jayant K, Malvi SG, Siddiqi M, Michel A, Butt J, Sankaran S, Kannan TPRA, Varghese R, Divate U, Willhauck-Fleckenstein M, Waterboer T, Muller M, Sehr P, Kriplani A, Mishra G, Jadhav R, Thorat R, Tommasino M, Pillai MR, Sankaranarayanan R; Indian HPV vaccine study group. Are two doses of human papillomavirus vaccine sufficient for girls aged 15-18 years? Results from a cohort study in India. Papillomavirus Res. 2018 Jun;5:163-171. doi: 10.1016/j.pvr.2018.03.008. Epub 2018 Mar 22. PMID 29578097
- [Result] Basu P, Muwonge R, Bhatla N, Nene BM, Joshi S, Esmy PO, Poli URR, Joshi G, Verma Y, Zomawia E, Shastri SS, Pimple S, Anantharaman D, Prabhu PR, Hingmire S, Sauvaget C, Lucas E, Pawlita M, Gheit T, Jayant K, Malvi SG, Siddiqi M, Michel A, Butt J, Sankaran S, Rameshwari Ammal Kannan TP, Varghese R, Divate U, Willhauck-Fleckenstein M, Waterboer T, Muller M, Sehr P, Vashist S, Mishra G, Jadhav R, Thorat R, Tommasino M, Pillai MR, Sankaranarayanan R; Indian HPV vaccine study group. Two-dose recommendation for Human Papillomavirus vaccine can be extended up to 18 years - updated evidence from Indian follow-up cohort study. Papillomavirus Res. 2019 Jun;7:75-81. doi: 10.1016/j.pvr.2019.01.004. Epub 2019 Jan 31. PMID 30711698
- [Result] Muwonge R, Basu P, Gheit T, Anantharaman D, Verma Y, Bhatla N, Joshi S, Esmy PO, Poli URR, Shah A, Zomawia E, Shastri SS, Pimple S, Prabhu PR, Hingmire S, Chiwate A, Sauvaget C, Lucas E, Malvi SG, Siddiqi M, Sankaran S, Kannan TPRA, Varghese R, Divate U, Vashist S, Mishra G, Jadhav R, Tommasino M, Pillai MR, Sankaranarayanan R, Jayant K; Indian HPV vaccine study group. Acquisition, prevalence and clearance of type-specific human papillomavirus infections in young sexually active Indian women: A community-based multicentric cohort study. PLoS One. 2020 Dec 29;15(12):e0244242. doi: 10.1371/journal.pone.0244242. eCollection 2020. PMID 33373380
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3-dose | 2-dose | 2 Doses by Default | Single-dose | Unvaccinated
Started | 4348 | 4979 | 3452 | 4950 | 5000
Completed | 4348 | 4979 | 3452 | 4950 | 4646
Not Completed | 0 | 0 | 0 | 0 | 354
Not completed — Ongoing enrollment | 0 | 0 | 0 | 0 | 354

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3-dose | 2-dose | 2 Doses by Default | Single-dose | Unvaccinated | Total
Number analyzed (Participants) | 4348 | 4979 | 3452 | 4950 | 4646 | 22375
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (2.3) | 13.6 (2.3) | 13.7 (2.4) | 13.7 (2.4) | 24.1 (2.9) | 15.8 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4348 | 4979 | 3452 | 4950 | 4646 | 22375
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Enrolment [Count of Participants; unit: Participants] | 4348 | 4979 | 3452 | 4950 | 4646 | 22375

OUTCOME MEASURES:

1. Primary Outcome: Median Florescent Intensities (MFI) of the Total Antibodies to Vaccine-included HPV Types (16/18/6/11) at Different Time Points
Description: Samples were treated with EDTA and analysed with Luminex (Austin, TX, USA) based multiplex serology to assess the concentration of binding antibodies against the major capsid protein L1 as mean median fluorescence intensity (MFI). MFI values as a measure of antibody concentration quantified by use of HPV multiplex serology are directly comparable with optical densities measured with ELISA.
Time Frame: Month 7 (for 3-dose and 2-dose groups), 12 (for 2 doses by default and single-dose groups), 18, 36, 48
Population: Data used for this outcome are from a subset of participants that had their immunogeneicity samples tested in the laboratory. We are indicating the total of HPV 16 L1 antibodies of the HPV 16 L1 antiboties at month 7 for the 3-dose and 2-dose groups and at month 12 for the 2 doses by default and single-dose groups. No immunogeneity data was collected from the unvaccinated cohort as it was recruited adhoc to assess the HPV infections and CIN endpoints.
Measure: Geometric Mean (95% Confidence Interval); unit: median flow intensities
Arm/Group | 3-dose | 2-dose | 2 Doses by Default | Single-dose | Unvaccinated
Number analyzed (Participants) | 308 | 317 | 471 | 528 | 0
median flow intensities | 5460 [5195 to 5738] | 6125 [5785 to 6485] | 437 [398 to 480] | 106 [96 to 116] |
Statistical Analysis 1: Comparison: 3-dose vs 2-dose vs 2 Doses by Default vs Single-dose; Test type: Non-Inferiority — To test for non-inferiority of antibody concentrations in different dose groups, log-transformed mean MFIs in linear regression models were used to obtain MFI ratios and their corresponding 95% confidence intervals (CIs). Antibody titres at months 0, 7, 12, 36 and 48 were compared and non-inferiority was inferred when the lower bound of the confidence interval of the ratio of the immunogenicity measures exceeded 0.5; Regression, Linear; Risk Ratio (RR) = 0.5 — The lower bound of the 95% CI ratio of immunogeneicity measures was used instead. No p-values were estimated

2. Primary Outcome: Frequency of Persistent HPV 16/18/6/11 Infection.
Description: The first cervical cell samples were collected from women 18 months after married or 6 months after the first delivery. After that, 3 extra annual collections were obtained. The HPV genotyping method involved HPV-type-specific E7 PCR bead-based multiplex genotyping. The multiplex HPV-type-specific E7 PCR uses HPV type-specific primers targeting the E7 region for the detection of 19 high-risk or probable high-risk HPV types (16, 18, 26, 31, 33, 35, 39, 45, 51, 52, 53, 56, 58, 59, 66, 68a, 68b, 70, 73, and 82), and two low-risk HPV types (6 and 11), with detection limits ranging from ten to 1000 copies of the viral genome.
Time Frame: From date of marriage through to 7 years of follow-up
Population: Participants with at least two cervical cell sample collections, that were collected at least 10 months apart.
Measure: Number; unit: Infections
Arm/Group | 3-dose | 2-dose | 2 Doses by Default | Single-dose | Unvaccinated
Number analyzed (Participants) | 1460 | 1452 | 1626 | 2135 | 1265
Infections | 1 | 1 | 4 | 1 | 32
Statistical Analysis 1: Comparison: 3-dose vs 2-dose vs 2 Doses by Default vs Single-dose vs Unvaccinated; Test type: Superiority; Vaccine efficacy = 95

3. Primary Outcome: Frequency of HPV 16/18-associated Precancerous Lesions and Cancer.
Description: Pathology Panel diagnosis of: CIN 2, CIN 3 (including squamous carcinoma in situ), adenocarcinoma in situ, invasive squamous cervical carcinoma, or invasive adenocarcinoma of the cervix and detection of HPV 16 and/or HPV 18 by PCR in the same biopsy tissue sample.
Time Frame: Cervical samples for HPV testing collected from married participants at the age of 25 and at 5 years after the first screen
Reporting Status: Not Posted, anticipated posting 2027-07

4. Secondary Outcome: Frequency of Infection by Other Non-targeted High-risk HPV Types.
Description: The HPV genotyping method involved HPV-type-specific E7 PCR bead-based multiplex genotyping. The multiplex HPV-type-specific E7 PCR uses HPV type-specific primers targeting the E7 region for the detection of 19 high-risk or probable high-risk HPV types (16, 18, 26, 31, 33, 35, 39, 45, 51, 52, 53, 56, 58, 59, 66, 68a, 68b, 70, 73, and 82), and two low-risk HPV types (6 and 11), with detection limits ranging from ten to 1000 copies of the viral genome.
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2027-07

5. Secondary Outcome: Frequency of Cervical Neoplasia Associated With Non-included HPV Types.
Description: Pathology Panel diagnosis of: CIN 2, CIN 3 (including squamous carcinoma in situ), adenocarcinoma in situ, invasive squamous cervical carcinoma, or invasive adenocarcinoma of the cervix and detection of other non vaccine included HPV types by PCR in the same biopsy tissue sample.
Time Frame: 15 years from the base-line date
Reporting Status: Not Posted, anticipated posting 2027-07

ADVERSE EVENTS:
Time Frame: 7 years
Arm/Group | 3-dose | 2-dose | 2 Doses by Default | Single-dose | Unvaccinated
All-Cause Mortality (participants affected / at risk) | 30/4348 | 22/4979 | 38/3452 | 45/4950 | 9/4646
Serious Adverse Events (participants affected / at risk) | 125/4348 | 135/4979 | 292/3452 | 356/4950 | 0/4646
Other Adverse Events (participants affected / at risk) | 637/4348 | 614/4979 | 614/3452 | 296/4950 | 0/4646
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3-dose (N=4348) | 2-dose (N=4979) | 2 Doses by Default (N=3452) | Single-dose (N=4950) | Unvaccinated (N=4646)
Hospitalization (Investigations) | 14 (14) | 26 (26) | 20 (20) | 26 (26) | 0 (0) — Hospitalized for illnesses
Abortion/Gynecological conditions (Pregnancy, puerperium and perinatal conditions) | 94 (94) | 92 (92) | 214 (214) | 239 (239) | 0 (0) — Spontaneous/ elective abortions; Gynecological Conditions
Preterm delivery (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 11 (11) | 28 (28) | 40 (40) | 0 (0) — Premature delivery/Congenital Anomaly
Neonatal death (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 6 (6) | 30 (30) | 51 (51) | 0 (0) — Neonatal Death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3-dose (N=4348) | 2-dose (N=4979) | 2 Doses by Default (N=3452) | Single-dose (N=4950) | Unvaccinated (N=4646)
Mild: Abdominal cramps (General disorders) | 5 (5) | 5 (5) | 2 (2) | 3 (3) | 0 (0)
Mild: Diarrhea (General disorders) | 5 (5) | 9 (9) | 3 (3) | 2 (2) | 0 (0)
Mild: Discomfort (General disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Mild: Dizziness (General disorders) | 18 (18) | 21 (21) | 22 (22) | 10 (10) | 0 (0)
Mild: Fainting (vaso vagal reaction) within 15 to 20 minutes of vaccine receipt (General disorders) | 4 (4) | 6 (6) | 0 (0) | 2 (2) | 0 (0)
Mild: Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mild: Injection site pain (General disorders) | 344 (344) | 341 (341) | 352 (352) | 137 (137) | 0 (0)
Mild: Joint stiffness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Mild: Low-grade fever (< 39°C sublingual) measurement) (General disorders) | 88 (88) | 80 (80) | 96 (96) | 76 (76) | 0 (0)
Mild: Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mild: headaches (General disorders) | 27 (27) | 18 (18) | 18 (18) | 8 (8) | 0 (0)
Mild: injection site swelling (General disorders) | 41 (41) | 26 (26) | 58 (58) | 22 (22) | 0 (0)
Mild: irritability (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mild: muscle pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mild: Muscle spasms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mild: Nausea (General disorders) | 15 (15) | 9 (9) | 6 (6) | 3 (3) | 0 (0)
Mild: Neck pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mild: Pain in extremity (General disorders) | 2 (2) | 5 (5) | 0 (0) | 6 (6) | 0 (0)
Mild: Rash (General disorders) | 0 (0) | 3 (3) | 8 (8) | 4 (4) | 0 (0)
Mild: Redness, mild tenderness or bruising around the injection site (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Mild: Sensation of heaviness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mild: Shoulder pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mild: Skin irritation (General disorders) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Mild: Other specify (General disorders) | 52 (52) | 53 (53) | 19 (19) | 10 (10) | 0 (0)
Moderate: Allergic reaction [Characterized by one or more of the following: (1) skin manifestations (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Moderate: Allergic skin reactions (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Moderate: Facial edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Moderate: High fevers sometimes associated with seizures (> 39° C) (General disorders) | 3 (3) | 5 (5) | 9 (9) | 3 (3) | 0 (0)
Moderate: Larger reactions (> 2 cm) around the injection site (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Moderate: Temporary joint pain or swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Moderate: Other specify (General disorders) | 21 (21) | 17 (17) | 7 (7) | 7 (7) | 0 (0)

LIMITATIONS AND CAVEATS:
Because of the suspension of all HPV vaccine studies for reasons not related to this trial, the study was able to recruit 17729 of the originally planned 20000 participants some of who received less than the originally planned vaccine dose schedule.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No